CLINICAL TRIAL: NCT01373593
Title: Ultrasound Guided Blocks of the Iliohypogastric and Ilioinguinal Nerves in Persistent Postherniorrhaphy Pain Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Joakim Bischoff, Rigshospitalet, Blegdamsvej 9, 2100 Copenhagen, Danmark
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: H-1-2010-116
Record Dates: First submitted 2011-06-08; First posted 2011-06-15 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2011-01

CONDITIONS: Pain
Keywords: persistent postherniorrhaphy pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- lidocaine (Experimental): lidocaine block
  Interventions: Drug: lidocaine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lidocaine
  Arms: lidocaine
Drug: Placebo
  Arms: Placebo

SUMMARY:
In this controlled study the investigators will examine the analgesic and sensory effects of ultrasound-guided blocks of the iliohypogastric and ilioinguinal nerves with lidocaine in persistent postherniorrhaphy pain patients.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years with severe postherniorrhaphy pain (numerical rating scale [NRS] > 6) for more than 6 month

Exclusion Criteria:

* known amide local anesthetic drug allergy
* recurrent hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
changes (lidocaine vs. placebo) in pain perception, sensory mapping and QST compared to pre-block values. | 20 minutes after the block

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Bischoff JM, Koscielniak-Nielsen ZJ, Kehlet H, Werner MU. Ultrasound-guided ilioinguinal/iliohypogastric nerve blocks for persistent inguinal postherniorrhaphy pain: a randomized, double-blind, placebo-controlled, crossover trial. Anesth Analg. 2012 Jun;114(6):1323-9. doi: 10.1213/ANE.0b013e31824d6168. Epub 2012 Mar 30. PMID 22467891